CLINICAL TRIAL: NCT03061955
Title: Safety and Efficacy of Concurrent Administration of Influenza Vaccine in Patients Undergoing Anti-PD-1 Immunotherapy (Nivolumab, Pembrolizumab)
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 6443
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2019-07

CONDITIONS: Influenza Virus Vaccine Adverse Reaction (Disorder); Influenza; Malignancy
MeSH Terms: conditions — Influenza, Human; Neoplasms | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: influenza vaccination — administration of influenza vaccination

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of concurrent administration of influenza vaccine in patients receiving anti-PD1 immunotherapy (nivolumab or pembrolizumab). This will be a prospective observational study, aiming to assess patient tolerance of treatment, adverse events (incidence, grade, need for hospitalization), incidence of influenza infections, and seroconversion rates.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Currently receiving immunotherapy with anti-PD-1 agents (Nivolumab or Pembrolizumab)
* Have not received influenza vaccination prior to study entry date for the upcoming flu season 2016-2017
* No previous contraindication to receiving influenza vaccination
* Histologically proven cancer
* Expected lifetime of at least 12 weeks

Exclusion Criteria:

* Previous cancer
* Autoimmune disease or immunosuppressive treatments
* Corticosteroid treatment
* Those who have a potential indication to change chemotherapy treatment in 42 days following start of treatment
* History of clinically or virologically confirmed influenza infection in the previous six months
* Previous contraindication to receiving influenza vaccination
* Previous allergic/adverse reaction with influenza vaccination
* Have received influenza vaccination prior to study entry date for upcoming 2016-2017 flu season
* Positive anti influenza antibody titers as determined by the baseline blood determination (day 0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older or are receiving either nivolumab or pembrolizumab who have no yet received the influenza vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Number of participants with confirmed influenza infection as assessed by influenza rapid antigen A and B testing, nose swab. | October 1st 2016 to March 31st 2017
  participants with confirmed influenza infection as assessed by influenza rapid antigen A and B testing, nose swab.

SECONDARY OUTCOMES:
Number of participants with adverse events and grading of adverse event as measured by the adverse events toxicity scale. | October 1st 2016 to March 31st 2017
  participants with adverse events
Number of participants requiring hospitalizations for adverse events or influenza infection. | October 1st 2016 to March 31st 2017
  participants requiring hospitalizations
Number of participants with seroconversion as assessed by influenza A and B IgM and IgG titers. | October 1st 2016 to March 31st 2017
  participants with seroconversion

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kunisaki KM, Janoff EN. Influenza in immunosuppressed populations: a review of infection frequency, morbidity, mortality, and vaccine responses. Lancet Infect Dis. 2009 Aug;9(8):493-504. doi: 10.1016/S1473-3099(09)70175-6. PMID 19628174
- [Background] Mariotti J, Spina F, Carniti C, Anselmi G, Lucini D, Vendramin A, Pregliasco F, Corradini P. Long-term patterns of humoral and cellular response after vaccination against influenza A (H1N1) in patients with hematologic malignancies. Eur J Haematol. 2012 Aug;89(2):111-9. doi: 10.1111/j.1600-0609.2012.01793.x. Epub 2012 May 31. PMID 22540245
- [Background] Pollyea DA, Brown JM, Horning SJ. Utility of influenza vaccination for oncology patients. J Clin Oncol. 2010 May 10;28(14):2481-90. doi: 10.1200/JCO.2009.26.6908. Epub 2010 Apr 12. PMID 20385981
- [Background] Preventing Infections in Cancer Patients. 2015. (Accessed June 22, 2016, at https://www.cdc.gov/cancer/flu/.)
- [Background] Rousseau B, Loulergue P, Mir O, Krivine A, Kotti S, Viel E, Simon T, de Gramont A, Goldwasser F, Launay O, Tournigand C. Immunogenicity and safety of the influenza A H1N1v 2009 vaccine in cancer patients treated with cytotoxic chemotherapy and/or targeted therapy: the VACANCE study. Ann Oncol. 2012 Feb;23(2):450-7. doi: 10.1093/annonc/mdr141. Epub 2011 May 16. PMID 21576285
- [Background] Mulder SF, Jacobs JF, Olde Nordkamp MA, Galama JM, Desar IM, Torensma R, Teerenstra S, Mulders PF, Vissers KC, Punt CJ, de Vries IJ, van Herpen CM. Cancer patients treated with sunitinib or sorafenib have sufficient antibody and cellular immune responses to warrant influenza vaccination. Clin Cancer Res. 2011 Jul 1;17(13):4541-9. doi: 10.1158/1078-0432.CCR-11-0253. Epub 2011 Jun 28. PMID 21712444
- [Background] Monkman K, Mahony J, Lazo-Langner A, Chin-Yee BH, Minuk LA. The pandemic H1N1 influenza vaccine results in low rates of seroconversion for patients with hematological malignancies. Leuk Lymphoma. 2011 Sep;52(9):1736-41. doi: 10.3109/10428194.2011.584003. Epub 2011 Jun 12. PMID 21663502
- [Background] Yri OE, Torfoss D, Hungnes O, Tierens A, Waalen K, Nordoy T, Dudman S, Kilander A, Wader KF, Ostenstad B, Ekanger R, Meyer P, Kolstad A. Rituximab blocks protective serologic response to influenza A (H1N1) 2009 vaccination in lymphoma patients during or within 6 months after treatment. Blood. 2011 Dec 22;118(26):6769-71. doi: 10.1182/blood-2011-08-372649. Epub 2011 Nov 4. PMID 22058114
- [Background] Weber JS, Hamid O, Chasalow SD, Wu DY, Parker SM, Galbraith S, Gnjatic S, Berman D. Ipilimumab increases activated T cells and enhances humoral immunity in patients with advanced melanoma. J Immunother. 2012 Jan;35(1):89-97. doi: 10.1097/CJI.0b013e31823aa41c. PMID 22130166